CLINICAL TRIAL: NCT04010045
Title: REvascularization RateS and Clinical OUtcomes With DABRA Laser. A Long-Term 2-year Study (RESULTS)
Brief Title: REvascularization RateS and Clinical OUtcomes With DABRA Laser. A Long-Term 2-year Study
Acronym: RESULTS
Status: Terminated | Type: Observational
Why Stopped: Sponsor stopped the study for business reasons as site recruitment and subject enrollment have not met expectations.
Sponsor: Ra Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: RMS-104
Record Dates: First submitted 2019-06-04; First posted 2019-07-08 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Artery Disease
Keywords: lower extremity PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Endovascular Treatment of PAD — PAD endovascular treatment using the DABRA Laser System + other FDA cleared/ approved devices for the treatment of PAD.
  Other Names: PAD endovascular treatment using the DABRA Laser System

SUMMARY:
This is an observational study of the DABRA Laser System and other medical devices intended for endovascular treatment of peripheral artery disease.

DETAILED DESCRIPTION:
This is an observational, prospective, consecutively enrolled, single-arm, multi-site registry of the use of the DABRA Laser System and other medical devices intended for endovascular treatment of peripheral artery disease.

This study covers the use of endovascular devices including the DABRA Laser System and other devices commercially used in the United States for the treatment of lower extremity PAD.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age ≥ 22 years.
* Participant presents with a Rutherford category of 2 to 6.
* Participant has at least one peripheral lesion, ≤ 140mm, in a native vessel that is treated successfully with DABRA Laser System.
* Participant is able and willing to be anti-coagulated.
* Ability and willingness of participant to give written informed consent and comply with follow-up.

Exclusion Criteria:

* Pregnant, breastfeeding, planning to become pregnant - If women of reproductive capability will be enrolled, status will be assessed via pregnancy testing. Subject must agree to use effective birth control measures for duration of study. Pregnancy during study must be reported immediately.
* Endovascular interventions within 90 days prior to study enrollment (on leg to be treated).
* Participation in another cardiovascular or peripheral vascular study that might, in the judgement of the Investigator, affect the results of the study.
* Disorders or allergies precluding use of radiographic contrast including renal insufficiency severe enough to contraindicate use of radiographic contrast.
* Inability or unwillingness of the patient to comply with study examinations.
* Necrosis necessitating major amputation.
* Subject has an anticipated life span of less than one (1) year.
* Medically non-compliant subjects, based on Investigator judgment (e.g., subject is non-compliant in following medical advice regarding blood pressure medication, cholesterol medication, and/or maintenance of healthy blood sugar levels).
* No run-off vessel is present when treating above the knee. A run-off vessel is required when treating above the knee, however, it is not required when treating below the knee.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is patients presenting with symptoms of peripheral artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Vessel Patency | 24 months
  Patency of the target lesion at 24 months, as determined by duplex ultrasound.

SECONDARY OUTCOMES:
Serious Adverse Events | 1 day, 6 months, 12 months, 18 months, and 24 months
  Tabulation of serious adverse events at 1 day, 6 months, 12 months, 18 months, and 24 months
Vessel Patency | 6 months, 12 months, and 18 months
  Patency of the target lesion at 6 months, 12 months, and 18 months, as determined by duplex ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Jami Miller, Study Director — Ra Medical Systems
Locations (1):
- NAADI Healthcare, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No